CLINICAL TRIAL: NCT02315040
Title: Testing the Effect of Intrauterine Slow Release Insemination (SRI) on the Pregnancy Rate in Women Designated for Standard Intrauterine Insemination (IUI)
Brief Title: EVIE-Study: Slow Release Insemination Versus Standard Intrauterine Insemination Study
Acronym: EVIE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Reproductive Sciences Ltd. (Unknown)
Responsible Party: Principal Investigator, Maximilian Franz, M.D., MD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: V1.2
Record Dates: First submitted 2014-10-19; First posted 2014-12-11 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-01

CONDITIONS: Insemination
Keywords: Intrauterine insemination (IUI); Insemination method; Slow release insemination (SRI); EVIE; Pregnancy rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IUI (Active Comparator): standard intrauterine insemination method
  Interventions: Other: Standard Intrauterine Insemination
- EVIE (Experimental): Slow release insemination method (SRI)
  Interventions: Device: EVIE

INTERVENTIONS:
Device: EVIE — EVIE is a small, mechanical, single use pump that mimics natural fertilization by introducing sperm into the uterus over a period of 4 hours, rather than all at once as in conventional IUI
  Other Names: Slow Release Insemination (SRI)
  Arms: EVIE
Other: Standard Intrauterine Insemination — standard intrauterine insemination procedure
  Other Names: IUI
  Arms: IUI

SUMMARY:
Overall Study Design and Plan Description

* The study will be conducted on women with fertility difficulties who are designated for intrauterine insemination treatment (IUI). The research sample size is 137 treatment cycles per group (total of 274 treatment cycles). The women will be randomly divided into two groups. Some will undergo the standard bolus IUI treatment and others will be treated with the EVIE Slow Release Insemination method (SRI). Women who fail to conceive in the first treatment will next receive the alternative treatment. This means that a woman treated with the IUI method who does not become pregnant will then be treated with SRI, and vice versa (crossover method). The study will include women treated with Clomiphene Citrate or with other Gonadotropin-based treatment. Every couple treated will undergo at least 2 insemination cycles (unless pregnancy has already been achieved).
* Before beginning the hormone treatment, each couple will have the trial procedure explained to them. This explanation will include all the detailed information and instruction about the IUI and the Slow Release Insemination methods. A Patient Information Sheet will be available to them.
* Preparation of the spermatozoa for intra uterine insemination will be identical to the method performed currently before IUI.

Approximately two weeks after the insemination treatment, a blood sample will be taken from the woman to check for Beta hCG levels to indicate pregnancy.

Hypothesis:

SRI leads to higher pregnancy rates compared to standard IUI

Primary endpoint:

• Pregnancy rate Effect of controlled Intra-uterine slow release insemination on the pregnancy rate of women designated for intra uterine insemination in comparison to the accepted IUI method.

ELIGIBILITY:
Inclusion Criteria:

1. Women with primary or secondary infertility after 6 months of unprotected intercourse who are candidates for IUI
2. Age of the woman - 20 to 40 years old
3. Normal uterus x-ray (HSG) or Chromotubation to determine tubal patency
4. Women with infertility on a background of non-ovulation
5. Infertility on a background of a male problem (over 10 million/ml motile sperm cells per sample)
6. Infertility on a background of unexplained cause
7. Same sex patient / single patient
8. Signed informed consent

Exclusion Criteria:

1. Woman under the age of 20 or over the age of 40 years
2. Female infertility on mechanical background affecting the uterus or Fallopian tubes
3. Infertility on male background of medium to very low level of spermatozoa - less than 10 million/ml motile sperm cells per sample
4. Men and women who are opposed to the random spermatozoa insemination method
5. Participants who are not willing to sign the Consent Form
6. BMI >30

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | average time frame: 2 weeks after insemination
  ß-HCG examination in urine or serum

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian B Franz, MD, Study Chair — Medical University of Vienna; Christian Egarter, MD, Prof., Principal Investigator — Medical University of Vienna; Julian Marschalek, MD, Study Chair — Medical University of Vienna
Locations (12):
- Austria (3):
  - Das Kinderwunsch Institut Schenk GmbH, Dobl
  - Dept. Obstetrics and Gynaecology, Medical University of Vienna, Vienna
  - Kinderwunschzentrum der Goldenes Kreuz Privatklinik, Vienna
- CRES Hopital Natecia, Lyon, France
- Germany (6):
  - Dept. Obstetrics and Gynaekology, Medical Faculty of Aachen, Aachen, Westfalen
  - Klinikum der Johann Wolfgang-Goethe-Universität Klinik für Frauenheilkunde und Geburtshilfe, Frankfurt am Main
  - Frauenärztliche Gemeinschaftspraxis Dr. Maarten R. van Santen; KriegsstraBe 216, Karlsruhe
  - LMU, Klinikum der Universität München Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Munich
  - Kinderwunsch Centrum München Pasing, Munich
  - Kinderwunschzentrum München Bogenhausen, Munich
- United Kingdom (2):
  - Fertility Fusion/Withington Hospital, Withington, Lancashire
  - Centre for Reproductive and Genetic Health - Eastman Dental Hospital, London, UK

REFERENCES:
- [Background] Muharib NS, Abdel Gadir A, Shaw RW. Slow release intrauterine insemination versus the bolus technique in the treatment of women with cervical mucus hostility. Hum Reprod. 1992 Feb;7(2):227-9. doi: 10.1093/oxfordjournals.humrep.a137622. PMID 1577936